CLINICAL TRIAL: NCT01783782
Title: SMALL BOWEL CLEANSING FOR CAPSULE ENDOSCOPY IN PEDIATRIC PATIENTS: A PROSPECTIVE RANDOMIZED SINGLE-BLINDED STUDY
Brief Title: Small Bowel Cleansing for Capsule Endoscopy in Pediatric Patients
Acronym: PREP-CE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CLEANSING FOR PED-CE
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2005-11

CONDITIONS: Capsule Endoscopy
Keywords: Capsule Endoscopy; colon cleansing; children; age 2 -18 years
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- DIET (Experimental): Group A followed the standard regime consisting of a clear liquid diet for 12 hours on the day before CE, followed by an overnight fast.
  Interventions: Behavioral: DIET
- HIGH PEG (Experimental): Group B received a high volume regime consisting of a 50 mL/Kg (up to 2 Lt/die) of polyethylene glycol 4000 solution with simethicon solution the evening before the examination, followed always by an overnight fast.
  Interventions: Drug: polyethylene glycol 4000 solution with simethicon
- LOW PEG (Experimental): Group C, defined as a low volume regime, received 25 mL/Kg (up to 1Lt/die) of polyethylene glycol 4000 solution with simethicon solution the evening before the examination, followed by an overnight fast.
  Interventions: Drug: polyethylene glycol 4000 solution with simethicon
- SIMETHICONE (Experimental): Group D received 20 mL oral simethicone (Panamir, DMG, Italy, containing 40 mg simethicone in 1mL emulsion) and 200mL water 30 minutes before capsule ingestion.
  Interventions: Drug: simethicon
- SIMETH+PEG (Experimental): Group E received 25 mL/Kg (up to 1 Lt/die) of polyethylene glycol 4000 solution with simethicon solution followed by an overnight fast plus 20mL oral simethicone and 200mL water 30 minutes before capsule ingestion.
  Interventions: Drug: polyethylene glycol 4000 solution with simethicon; Drug: simethicon

INTERVENTIONS:
Behavioral: DIET — clear liquid diet for 12 hours on the day before CE, followed by an overnight fast
  Arms: DIET
Drug: polyethylene glycol 4000 solution with simethicon — patients received a high volume regime consisting of a 50 mL/Kg (up to 2 Lt/die) of PEG solution the evening before the examination, followed always by an overnight fast
  Other Names: selg-esse
  Arms: HIGH PEG; LOW PEG; SIMETH+PEG
Drug: simethicon — Patients received 20 mL oral simethicone (Panamir, DMG, Italy, containing 40 mg simethicone in 1mL emulsion) and 200mL water 30 minutes before capsule ingestion
  Other Names: Panamir V
  Arms: SIMETH+PEG; SIMETHICONE

SUMMARY:
The primary aim of this prospective, randomized and controlled study was to evaluate the effect of five bowel preparation regimens on small-bowel cleansing in a pediatric population. The secondary endpoints were to evaluate the safety and the effects of preparation on diagnostic yield of CE.

DETAILED DESCRIPTION:
Capsule endoscopy (CE) is a well-known, non-invasive, diagnostic tool to evaluate small bowel diseases in adults and children. Unfortunately, because CE does not have functions which allow suctioning of fluid or washing the small bowel mucosa during the examination, its diagnostic yield can be limited by presence of debris, biliary secretion, bubbles and blood in the gut lumen that may hide relevant findings especially in the distal small bowel. In addition, CE sometimes fails to reach the cecum within the battery life of the capsule, resulting in a failure to visualize the distal small intestine. However, in children this problem is less frequent for the increased intestinal motility, which reduces the transit time of the capsule.

It was believed that cleaning the small intestine prior to examination would improve mucosal visibility during the endoscopy and, as a result, the diagnostic yield of the technique. Therefore, proposals were put forward based on preparations for other types of explorations, such as colonoscopies (2).

Some authors have already studied in adults the effect of bowel preparation on small-bowel visualization using different agents; the results of the published series are contradictory. To date, while there is evidence for a benefit from bowel preparation for CE, there is so far no consensus on an optimal preparation regimen. In addition, in children there are not studies on this topic. Therefore, overnight fasting before the examination still remains the proposed preparation for capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Small Bowel capsule endoscopy in our Institution between 2 and 18 years of age were recruited for this study.

Exclusion Criteria:

* intestinal obstruction,
* suspicious impaired intestinal motility,
* history of gastrointestinal surgery

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-11; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy | During the performance of capsule endoscopy
  Preparation efficacy was evaluated by the blinded endoscopist according to a visibility score.
  There is no standardized or validated scoring system for the quality of small-bowel cleanliness. The visibility of the mucosal surface was assessed as the percentage of visualized bowel surface area as follows: 1: < 25%; 2: 25%-49%; 3: 50%-74%; 4: 75%-89%; 5: > 90%.

SECONDARY OUTCOMES:
Efficacy | during the reading capsule endoscopy
  the number of positive findings and the overall diagnostic yield.
  A positive finding was defined as the presence of a visible finding, whether incidental or clinically relevant. A positive yield at CE was assumed if the visible finding was considered relevant to the indication for CE. Where appropriate, this was confirmed by further evaluation (repeated upper-GI or lower-GI endoscopy, single-balloon enteroscopy (SBE), laparotomy, or cross-sectional imaging).
Safety | 4 days
  Adverse events were assessed on the day of capsule endoscopy by direct questioning and by telephone interview 48-96 hours after capsule endoscopy.
clinical tolerabiity | On the morning of colonoscopy, immediately before the procedure
  Tolerability assessment was based on the recording of occurrence and severity of GI symptoms such as nausea, bloating, abdominal, pain/cramps and anal discomfort.
  All patients were tested with a questionnaire, based on a numerical scale between 0 and 10 (with 10 being no burden at all and 0 indicating an intolerable procedure), about the impact of the bowel preparation (Van Tuyl Endoscopy 2007) and their level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Pediatrics, Sapienza - University of Rome, Rome, Rome, Italy